CLINICAL TRIAL: NCT05057416
Title: The Effect of Exercise Intensity on Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 119244
Record Dates: First submitted 2021-08-16; First posted 2021-09-27 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Exercise Adherence; Physical Activity Enjoyment; Cardiometabolic Health; Cardiovascular Health

STUDY DESIGN:
Intervention Model Description: This study will be include females aged 20-49, 3 exercise conditions analyzed for exercise enjoyment and adherence. It will involve 30 women assigned randomly to one of three exercise groups with a specific exercise protocol with various intensities. The study will be 8 weeks in duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (HIIT) Protocol (Experimental): Participants in the HIIT group will start with a 2.5-minute warm-up at about 30% VO2 max. The participants will then complete 3 running bouts at 80-90% VO2 max. Each running bout will be separated by 2 minutes of active rest where the participants will walk at 50% VO2 max. The total exercise time of this protocol will be 15 minutes. Finally, the participants will finish with a 2.5 min cool-down where they will walk at a light intensity of 30% VO2 max, for a total exercise duration of 20 minutes.
  Interventions: Behavioral: Exercise Adherence
- Sprint Interval Training (SIT) Protocol (Experimental): Participants in the Sprint Interval Training group will perform a 2.5-minute warm up at a VO2 max of 30%. Next, the participants will perform 6 all-out sprints at 150-200% of VO2 max, separated by 2-minute active rests at 50% VO2 max. The total exercise time of the SIT protocol is about 14 minutes. Finally, the participants will perform a walking cool-down of 3.5 minutes at 30% VO2 max, for a total exercise duration of 20 minutes.
  Interventions: Behavioral: Exercise Adherence
- Moderate Intensity Continuous Training (MICT)Protocol (Experimental): Participants in the Moderate Intensity Continuous Training group will first be warming up for 2.5 minutes at a VO2 max of 30%. After the warm up, participants will be running for 15 minutes at 45-60% of VO2 max. Finally, the participants will perform a 2.5-minute cool-down at 30% VO2 max, for a total exercise duration of 20 minutes.
  Interventions: Behavioral: Exercise Adherence

INTERVENTIONS:
Behavioral: Exercise Adherence — Our current study will compare three exercise groups which will all vary in intensity. Participants will be randomly assigned to one of the three groups. Two groups will be assigned to high intensity bouts of exercise with an active rest between, and one group will perform moderate intensity continuous training without resting. All groups will exercise for 20 minutes. Exercise adherence and it will be measured by a self-report online Google Document.

SUMMARY:
This study aims to advance the knowledge of a novel strategy of exercise to help people achieve the health benefits of exercise in less commitment time. As opposed to the traditionally recommended long periods (60 min) of moderate intensity exercise, this study will examine the effects of two exercise programs which consist of different intensities and repeated bouts of short intense exercise followed by rest periods. By incorporating short intense bouts of exercise, it may be possible that individuals enjoy this strategy of exercising more, which may influence them to continue to train in this way, increase their exercise levels in daily life and achieve exercise-related health benefits. Overall healthy women will be divided into a novel sprint interval training group or a high intensity interval training group or a traditional moderate intensity continuous training group. To evaluate the success of each training approach, a health-related quality of life questionnaire, one mile run test, weight, strength test and adherence to study requirements will be assessed over a 6-week period. The investigators hypothesize that the sprint interval training group will experience greatest strength measurements, will lose most body fat, have the greatest exercise benefits and will enjoy the novel training program more and will therefore adhere to the program more than the moderate continuous training group.

DETAILED DESCRIPTION:
Since the majority of the population is inactive, this study is being done to develop a better strategy that might encourage people to exercise more and improve their health. The current physical activity guidelines suggest that adults aged 18-64 should perform at least 150 minutes of moderate- to vigorous-intensity aerobic physical activity per week . However, 84% of the Canadian population is insufficiently active. The large percentage of inactive individuals may be due to the daunting expectation that individuals must exercise for long periods of time to achieve health benefits, and many individuals report not having enough time. However, studies have shown that exercising for short, repeated bouts of intense exercise resulted in improved cardiometabolic health to the same extent as traditional endurance training, despite lower exercise volume. One study found that the prescription for a higher frequency of exercise significantly increased the accumulation of exercise without a negative effect on adherence. Further, in another study, participants who performed short intense bouts of physical activity have shown greater adherence than participants who were performing traditional exercise, working at a moderate intensity for a prolonged exercise period (89% and 71%, respectively). None of the studies mentioned above examined time matched exercise groups and included varying intensities of exercise, and collected data through virtual means, mimicking the natural environment of participants. The investigators believe that the proposed study will address these concerns and therefore advance the knowledge of sprint interval training.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Participants must be between 20-49 years old
* Sedentary- completing less than 1 hour per week of leisure time physical activity over the prior 12 months and/or not meeting the CSEP guidelines of 150 minutes of moderate to vigorous physical activity per week
* Generally healthy males and females, no racial or gender bias.

Exclusion Criteria:

* Male
* Diagnosis of diabetes
* Taking glucose lowering medication
* Uncontrolled hypertension blood pressure >160/90
* History of heart disease
* Previous myocardial infarction or stroke
* Contraindications of exercise

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Estimated)
Dates: Start 2021-12-02 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Enjoyment | 8 weeks
  The enjoyment that participants experienced during the assigned intensity of exercise measured by the Physical Activity Enjoyment Scale (PAES).
Adherence to Exercise | 8 weeks
  Participants will report whether or not they have continued with the plan throughout the study duration through a weekly exercise diary.

SECONDARY OUTCOMES:
Exercise endurance | 8 weeks
  Participant cardiovascular endurance will be measured through a one-mile run test.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PHD, Principal Investigator — Western University
Locations (2):
- Canada (2):
  - Exercise Nutrition Laboratory (Western University), London, Ontario
  - Exercise Nutrition Laboratory, Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Plan to share IPD data in journals.
Supporting Information: Study Protocol, SAP
Time Frame: September 2022

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12211512/
- See also: Related Info — https://www.researchgate.net/publication/11176608_Adherence_to_exercise_prescriptions_Effects_of_prescribing_moderate_versus_higher_levels_of_intensity_and_frequency
- See also: Related Info — https://doi.org/10.1186/s12889-020-09234-y
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0154075